CLINICAL TRIAL: NCT03479359
Title: Learning Curve of Digital Rectal Examination for Prostate Cancer Among Internship
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zeng Shuxiong, Attending doctor in the Department of urology, Changhai Hospital
Other Study IDs: CH-Urology-DRE-001
Record Dates: First submitted 2018-03-08; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Prostatic Neoplasms; Digital Rectal Examination; Benign Prostatic Hyperplasia
Keywords: Prostate cancer; Benign Prostatic Hyperplasia; Digital Rectal Examination; Accuracy
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: In this group, internship are given the pathology outcome of each prostate biopsy regularly twice a month.
  Interventions: Behavioral: Routine review of DRE results by attending doctors
- Group 2: In this group, internship are not given the pathology outcome of each prostate biopsy.

INTERVENTIONS:
Behavioral: Routine review of DRE results by attending doctors — Let the internship regularly compare DRE result and the pathology outcome of prostate biopsy of each patient.
  Groups: Group 1

SUMMARY:
The investigators conduct this prospective study to investigate the learning curve of digital rectal examination (DRE) for prostate cancer among internship. The investigators want to know how many DRE are usually needed for internship to be performed in urological practice to obtain a stable DRE accuracy.

DETAILED DESCRIPTION:
Digital rectal examination (DRE) is a basic physical examination in routine practice in Urology. The DRE is a very important daily practice for screen prostate cancer, and each internship in Urology is required to perform this for patients suspected of prostate cancer or benign prostate hyperplasia. However, how many DRE are usually needed for a internship to perform so as to obtain a stable accuracy in daily practice is currently unknown. The investigators thus conduct this prospective trial to investigate the learning curve of DRE among internship.

ELIGIBILITY:
Inclusion Criteria:

* Internship just graduate from the medical school, and agree to attend the study.
* Internship have less than 5 DREs of prostate cancer.
* Patients of any age who are included for prostate biopsy are eligible, the indications for prostate biopsy are as follows: PSA>4ng/ml, fPSA/tPSA<0.16, with suspected palpable nodes in the prostate by DRE of attending doctor, suspected mass in prostate detected by ultrasound examination, magnetic resonance imaging, or computed tomography.

Exclusion Criteria:

* Internship who are not willing to attend the study.
* Internship stop doing DRE for continuously 3 months after entering the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All included internship are graduated from the Second Military Medical University and have already get the M.D. degree
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-02-26 (Estimated); Study Completion 2019-02-26 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of DRE performed by internship will be confirmed by prostate biopsy | One year
  To examine the sensitivity and specificity of the DRE performed by internship to reference standard of prostate biopsy in a prospective longitudinal cohort of around 700 participants who will undergo prostate biopsy due to suspect of prostate cancer. The investigators will investigate the sensitivity and specificity of DRE by different internship monthly.

SECONDARY OUTCOMES:
Sensitivity and specificity of DRE performed by internship with different training plan will be confirmed by prostate biopsy | One year
  To examine the sensitivity and specificity of the DRE performed by internship (group 1 with routinely review of pathologic outcome of prostate biopsy twice a month, and group 2 internship who are not told the results of prostate biopsy) to standard reference of prostate biopsy.
Sensitivity and specificity of DRE performed by internship will be compared to the results of fPSA/tPSA and MRI. | One year
  To compare the sensitivity and specificity of DRE to fPSA/tPSA and MRI (not any patients are required to have MRI examination of prostate, this will be determined at the discretion of attending doctor) to reference standard of prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanliang Xu, M.D., Ph.D, Principal Investigator — Second Military Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after the results of the study has been published. Related information will be given if request by email is agreed by the principle investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be shared after the results of the study has been published.

REFERENCES:
- [Background] Halpern JA, Oromendia C, Shoag JE, Mittal S, Cosiano MF, Ballman KV, Vickers AJ, Hu JC. Use of Digital Rectal Examination as an Adjunct to Prostate Specific Antigen in the Detection of Clinically Significant Prostate Cancer. J Urol. 2018 Apr;199(4):947-953. doi: 10.1016/j.juro.2017.10.021. Epub 2017 Oct 20. PMID 29061540
- [Background] Clements MB, Schmidt KM, Canfield SE, Gilbert SM, Khandelwal SR, Koontz BF, Lallas CD, Liauw S, Nguyen PL, Showalter TN, Trabulsi EJ, Cathro HP, Schenkman NS, Krupski TL. Creation of a Novel Digital Rectal Examination Evaluation Instrument to Teach and Assess Prostate Examination Proficiency. J Surg Educ. 2018 Mar-Apr;75(2):434-441. doi: 10.1016/j.jsurg.2017.08.012. Epub 2017 Oct 12. PMID 28923535